CLINICAL TRIAL: NCT00487344
Title: Comparison of Body Fat Reduction in Overweight and Obese Subjects Utilizing Personalized Low-Fat Meal Plans vs. Non-Personalized Low-Fat Meal Plans.
Brief Title: Research Study of Nutritional Methods to Reduce Body Fat Percentages in Overweight and Obese Populations
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Central FITT, Inc (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: CF-01-D-0001
Record Dates: First submitted 2007-06-15; First posted 2007-06-18 (Estimated); Last update posted 2007-07-03 (Estimated); Status verified 2007-05

CONDITIONS: Obesity
Keywords: medicaid; insurance; education; clinical; trial; healthcare; reimburse; pay; free; assist; study; oklahoma; edmond; Oklahoma City; diet; nutrition; weight loss; body; fat; obese; overweight; health; medical; therapy; meal plan; jenny craig; weight watcher; LA Weightloss; Bryan Attebery; Results; YMCA; UCO; OSU; OU; clinics; physicians; surgery; pills; financial; money
MeSH Terms: conditions — Obesity; Helping Behavior; Weight Loss; Platelet Glycoprotein IV Deficiency; Overweight

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Non-Personalized Meal Planning
Procedure: Personalized Meal Planning and Dietetic Consultation

SUMMARY:
The purpose of this study is to compare the use of personalized low-fat meal plans vs. non-personalized low-fat meal plans and the results in body fat reduction in overweight and obese subjects 25 to 45 years of age.

Compensation to Eligible Participants:

1. FREE Nutritional Services will be provided to eligible participants, which normally have a business value of between $165.00 and $195.00.
2. Each eligible participant will receive compensation for mileage directly related to this study up to 35 miles at the 2007 IRS Business Mileage Reimbursement Rate for medical purposes of $0.20 per mile. This compensation will be provided to each eligible participant in the form of a complimentary Wal-mart Gift Card in the amount of $7.00, contingent upon his or her completion in the study.

DETAILED DESCRIPTION:
Study Rationale: This experiment on the effect that the use of personalized low-fat meal plans has on body fat reduction is important for several reasons. First, the details of this research study may equip the public with knowledge to select quality nutrition programs for weight loss responsibly. Second, it may encourage the wellness and fitness community to reconsider the practice of providing clientele with non-personalized meal plans for weight loss, which are not usually designed by accredited dietetic professionals. Third, this study may benefit dietetic professionals by opening the lines of communication between the wellness community and the dietetic community regarding standards of care, and protecting the public by dispelling harmful and erroneous nutrition advice.

ELIGIBILITY:
Inclusion Criteria:

* Between 25 to 45 years of age
* Classified as overweight or obese with body mass index (BMI) measurement between 25 and 50
* Limited to minor chronic health

Exclusion Criteria:

* Individuals with the following health conditions:
* Food allergies
* Food intolerances
* Cancer
* Debilitating joint conditions such as Degenerative Joint Disease (DJD) and Degenerative Disk Disease (DDD)
* Diabetes Mellitus receiving insulin therapy
* Kidney problems
* Menopause
* Polycystic ovarian syndrome (PCOS)
* Currently pregnant or breast feeding
* Using diuretics, chromium, and/or diet pills
* Participants must:
* Live in the following Oklahoma Counties:
* Canadian, Cleveland, Logan, Lincoln, Oklahoma, and Pottawatomie
* Will to travel to Edmond and Oklahoma City, Oklahoma

Ages: 25 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Estimated)
Dates: Start 2007-06; Study Completion 2007-11 (Estimated)

PRIMARY OUTCOMES:
Pre and Post-Bioelectrical Impedance Body Fat Analysis | 2 months

CONTACTS AND LOCATIONS:
Overall Officials: Judith Brooks, Phd, Study Chair — Eastern Michigan University CHHS Thesis Committee; Anahita Mistry, PhD, Study Chair — Eastern Michigan University-CHHS Thesis Committee
Locations (1):
- Central FITT Inc, Edmond, Oklahoma, United States